CLINICAL TRIAL: NCT07127003
Title: Prospective, Randomized Clinical Trial for Immediate Lymphatic Reconstruction to Prevent Breast Cancer Related Lymphedema
Brief Title: ILR to Prevent BRCL_MCC 23608
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY007686
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer Lymphedema
Keywords: Axillary lymph node dissection; breast cancer; lymphedema
MeSH Terms: conditions — Breast Cancer Lymphedema; Breast Neoplasms; Lymphedema

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALND plus Immediate lymphatic reconstruction (Experimental): Undergo ILR during ALND surgery, where preserved lymphatic channels are connected to nearby veins to prevent lymphedema.
  Interventions: Procedure: Immediate Lymphatic Reconstruction
- ALND Alone (No Intervention): Will not receive ILR, but efforts will be made to preserve lymphatic channels during surgery.

INTERVENTIONS:
Procedure: Immediate Lymphatic Reconstruction — Preserved lymphatic channels are connected to nearby veins to prevent lymphedema during the axillary lymph node dissection.
  Arms: ALND plus Immediate lymphatic reconstruction

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of Immediate Lymphatic Reconstruction (ILR) in preventing breast cancer-related lymphedema (BCRL) in high-risk patients. It will also assess the safety and quality of life outcomes associated with the procedure. The main questions it aims to answer are:

Does ILR reduce the incidence of BCRL in patients undergoing axillary lymph node dissection (ALND)?

What are the patient-reported outcomes and quality of life differences between those who receive ILR and those who do not?

Participants will be identified as high-risk for developing BCRL through a multidisciplinary tumor board and referred to a specialized clinic for further evaluation. High-risk patients will undergo a series of screening tests, including bioimpedance spectroscopy (BIS), circumferential limb measurements, and infrared 3D perometry.

Participants will be randomly assigned to one of two groups:

Intervention Group (Study Arm A): Undergo ILR during ALND surgery, where preserved lymphatic channels are connected to nearby veins to prevent lymphedema.

Control Group (Study Arm B): Will not receive ILR, but efforts will be made to preserve lymphatic channels during surgery.

Patients will be blinded to their group assignment. Post-surgery, all participants will receive education from a certified lymphatic physical therapist.

At the 2-week postoperative visit, participants will be further randomized into two postoperative monitoring protocols:

BCRL Clinical Pathway: Patients will have regular follow-up visits every three months for two years, including repeat BIS, limb measurements, perometry, and quality of life questionnaires (LYMQOL and ULL-27).

Standard of Care: Patients will be monitored only if they experience BCRL symptoms or after two years from ALND.

The study will compare the outcomes of both groups, with a focus on the incidence of BCRL and patient quality of life, and will benchmark these results against published literature on breast cancer patients.

DETAILED DESCRIPTION:
This study will be a randomized control trial. As part of our multidisciplinary lymphedema clinic, patients at high-risk for developing BCRL will be recruited as a part of our randomized control trial. Enrollment will last for 12 months. The clinic team consists of the plastic surgeon, certified lymphedema therapist, clinical nurse, and nutritionist. High-risk patients will be identified in breast oncology weekly multidisciplinary tumor board, consisting of surgical oncology, medical oncology, radiation oncology, and radiology, and referred to our high-risk screening clinic.

High-risk patient screening consists of serial bilateral upper extremity bioimpedance spectroscopy (BIS), bilateral upper extremity circumferential limb girth measurements, and infrared 3D perometry. At this point, the study participants with be randomized into two arms: the intervention group (study arm A) will proceed with ILR, and the control group (study arm B) will not have ILR. Patients will be blinded to which arm they are randomly assigned.

During surgery, patients identified as requiring ALND due to axillary nodal burden will initially undergo RAM. This facilitates identification of fine lymphatic structures in the axilla. Through collaborative ALND performed simultaneously with a breast surgical oncologist, microvascular lymphatic and venous dissection is performed concurrently with nodal extirpation. Every effort will be made to preserve lymphatic channels not involved in nodal extirpation in patients randomized to group B.

For patients randomized to undergo ILR, the preserved lymphatic channels are matched with nearby branches of the axillary vein (most commonly the thoracoepigastric vein) to ensure a tension-free anastomosis.

On postoperative day one, patient education by the certified lymphatic physical therapist is done prior to discharge from the hospital to all patients. Following surgery, at the 2-week postoperative clinic visit, study patients will be again randomized to specific postoperative evaluation protocols: our established BCRL Clinical Pathway, or 2) via standard of care. Patients randomized to postoperative monitoring via the BRCL Clinical Pathway will be seen every three months postoperatively for 24 months. The group with the standard of care will only be seen if they experience symptoms of BCRL or are two years out from ALND. The decision for two years was decided to encompass when the risk for the development of BCRL peaks around 6-12 months after ALND. During these BCRL Clinical Pathway clinic visits, repeat BIS, circumferential limb measurements, and perometry are obtained. Patients are also asked to complete patient reported outcomes questionnaires, including LYMQOL (Lymphoedema Quality of Life) and ULL-27 (Upper Limb Lymphedema 27). The LYMQOL and ULL-27 questionnaires will be utilized to assess quality of life and patient reported symptoms of BCRL. LYMQOL covers four domains: symptoms, body image/appearance, function, and mood. ULL-27 investigates physical functioning, psychological, and social dimensions of quality of life with BCRL. Outcomes will be compared to published literature in breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients consenting for unilateral ALND [prior history of sentinel lymph node biopsy (SLNBx) allowed if <6 months from consent]
* Patients consenting for unilateral SLNBx with possible ALND, with a clinically or radiographically positive lymph node OR a high likelihood of ALND per the Breast Surgeon
* Identification of at least one transected lymphatic channel and at least one vein to be used for bypass at the time of ALND during surgery
* Female breast cancer patients 18-75 years of age (inclusive)

Exclusion Criteria:

* • Male breast cancer patients

  * Non-English speaking participants
  * Female breast cancer patients with axillary recurrence
  * Female breast cancer patients who have a history of ALND
  * Female patients requiring bilateral ALND for the treatment of their breast cancer
  * Female breast patients treated with SLNBx only
  * Primary lymphedema of the affected upper limb
  * Secondary lymphedema of the affected limb prior to the lymphadenectomy
  * Radiotherapy at the axilla before the study / surgery
  * Life expectancy < 2 years for any reason
  * Pregnancy or nursing
  * Substance abuse (such as alcohol or drug abuse) within 6 months prior to screening
  * Severe psychiatric disease
  * Distant metastases at the time of preoperative screening

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of BCRL at 24-month post follow up visit | 24 months Post ALND
  Efficacy of ILR will be measured by the incidence of BCRL at the 24 month post follow up visit

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Tampa General Hospital, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of South Florida, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD

REFERENCES:
- [Background] Gradishar WJ, Moran MS, Abraham J, Abramson V, Aft R, Agnese D, Allison KH, Anderson B, Burstein HJ, Chew H, Dang C, Elias AD, Giordano SH, Goetz MP, Goldstein LJ, Hurvitz SA, Jankowitz RC, Javid SH, Krishnamurthy J, Leitch AM, Lyons J, Mortimer J, Patel SA, Pierce LJ, Rosenberger LH, Rugo HS, Schneider B, Smith ML, Soliman H, Stringer-Reasor EM, Telli ML, Wei M, Wisinski KB, Young JS, Yeung K, Dwyer MA, Kumar R. NCCN Guidelines(R) Insights: Breast Cancer, Version 4.2023. J Natl Compr Canc Netw. 2023 Jun;21(6):594-608. doi: 10.6004/jnccn.2023.0031. PMID 37308117
- [Background] Tourani SS, Taylor GI, Ashton MW. Understanding the three-dimensional anatomy of the superficial lymphatics of the limbs. Plast Reconstr Surg. 2014 Nov;134(5):1065-1074. doi: 10.1097/PRS.0000000000000640. PMID 25347638